CLINICAL TRIAL: NCT01805466
Title: A New Cardiopulmonary By-pass System That Minimizes Haemodilution, Hemolysis and Systemic Inflammation. Effects on Organ Damage and Surgical Outcome
Brief Title: Effects on Organ Damage and Surgical Outcome of a New Cardiopulmonary Pass System (EVADO)
Acronym: EVADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-2009-1591573
Record Dates: First submitted 2013-02-26; First posted 2013-03-06 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: Extracorporeal Vacuum Assisted Device Optimised (EVADO)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVADO (Experimental): The E.V.A.D.O. system is made of the following components:
  * The ADMIRAL oxygenator, that requires low priming volumes (, has a limited contact surface and contains an accessory independent cardiotomy reservoir, allowing separation of pericardial suction blood.
  * The HARMONY Smart Suction System, which allows automatic regulation of a pumpless extracavity blood sucker, whose rates and pressures depend on whether suction is required for blood/air surfaces (skimming), or for fluids (pooled).
  * Paediatric circuits with 3/8" tubing for both arterial and venous lines.
  Interventions: Device: EVADO
- Conventional CPB (Active Comparator): conventional cardiopulmonary by-pass (CPB) system
  Interventions: Device: Conventional CPB

INTERVENTIONS:
Device: EVADO — EVADO (Extracorporeal Vacuum-Assisted Device Optimized) device enables separation of cardiotomy suction blood, which is stored in a separate reservoir, and, if re-infusion into the CPB circuit is required, this is performed only after selective filtering and by cell saver procedures. Moreover, by using a vacuum-assisted system for blood aspiration, EVADO allows complete elimination of roller pumps, therefore reducing the extent of mechanical cellular trauma. EVADO contains a phosphorylcholine-coated oxygenator, that confers superior biocompatibility. Finally, by requiring relatively limited priming volumes, it allows reducing haemodilution.
  Arms: EVADO
Device: Conventional CPB — conventional miniature cardiopulmonary bypass technique
  Arms: Conventional CPB

SUMMARY:
The primary purpose of this study is to assess the effects of the use of EVADO with respect to a conventional cardio-pulmonary bypass (CBP) system on surgical morbidity and mortality. As secondary aim this study wants to conduct appropriate laboratory investigations in order to detect the major biological mechanisms potentially responsible for the beneficial effects of the EVADO system on the coagulation cascade and inflammatory activation.

DETAILED DESCRIPTION:
The present study is designed as a prospective, multicentre, randomized, open label, controlled, 2-arm parallel group, superiority trial.

Participating centres are selected based on previous experience with the use of the EVADO system.

Patients elected to open heart surgery for a variety of cardiac conditions related to coronary, valvular or aortic disease or their combination in the participating centers will be screened.

This study as secondary aim wants to confirm the results of earlier investigation by a multicentre trial conducted on a larger population of patients undergoing a wide spectrum of open heart cardiac operations and either assess a number of cost-efficacy-efficiency indicators.

ELIGIBILITY:
Inclusion Criteria:

patients elected to undergo open heart surgery for a variety of cardiac conditions related to coronary, valvular or aortic disease or their combination and fulfilling the following additional criteria:

* Written informed consent
* Age 18-85 years

Exclusion Criteria:

* Severe renal or liver failure
* Uncompensated diabetes
* Autoimmune disease requiring immunosuppressant therapy
* Coagulation disorders
* Emergent or redo surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
composite of in-hospital mortality and clinical and outcome parameters recorded in the post-operative period | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The primary efficacy endpoint is the composite of in-hospital mortality, defined as death of any cause occurring before hospital discharge, myocardial infarction, stroke; severe renal failure; severe liver failure; severe cardio-respiratory failure; multiorgan failure; need for left ventricular support device; need for dialysis or ultrafiltration: post-operative bleeding; atrial fibrillation.

SECONDARY OUTCOMES:
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period: Myocardial infarction
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Stroke
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Severe renal failure (greater than 2-fold increase in creatinine levels)
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Multiorgan failure (MOF)
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Need for left ventricular support device (IABCP or similar)
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Need for dialysis or ultrafiltration
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Postoperative bleeding
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Atrial fibrillation
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Severe liver failure (greater than 2-fold increase in AST (aspartate aminotransferase), ALT (alanine aminotransferase) and y-GT (y-glutamyltransferase) levels)
Individual components of the primary end-point | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  outcome parameters recorded in the postoperative period:
  Severe cardio-respiratory failure

OTHER OUTCOMES:
Other pre-specified outcome measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  • Total duration of hospital admission [Time Frame: participants will be followed for the duration of hospital stay, an expected average of 2 weeks] [Designated as safety issue: Yes]
Other pre-specified outcome measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  • Duration of ICU stay
Other pre-specified outcome measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  • Time to extubation
Other pre-specified outcome measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  • Total postoperative blood loss and blood transfusion volume
Other pre-specified outcome measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  • Total hospitalization costs
Other pre-specified outcome measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  • Cost-efficiency assessment

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Nasso, MD, Principal Investigator — IRCCS San Raffaele Pisana
Locations (4):
- Italy (4):
  - Anthea Hospital, Bari
  - Maria Cecilia Hospital, Cotignola
  - Città di Lecce Hospital, Lecce
  - ICLAS Rapallo, Rapallo